CLINICAL TRIAL: NCT00190047
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Study To Evaluate The Effects Of DP-b99 On Neurologic Function And Disability In Subjects With Acute Ischemic Hemispheric Stroke
Brief Title: Effects Of DP-b99 On Neurological Function In Subjects With Acute Ischemic Hemispheric Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: D-Pharm Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ptcl-01213
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Brain Ischemia; Stroke; Cerebrovascular Disorders
Keywords: Cerebral Ischemia; Ischemic Brain Injury; Brain Infarction; Brain Ischemia
MeSH Terms: conditions — Brain Ischemia; Stroke; Cerebrovascular Disorders; Brain Infarction | interventions — DP-b99

INTERVENTIONS:
Drug: DP-b99

SUMMARY:
This study will examine if DP-b99 can improve neurological function (for example strength and coordination) in the 3 months after an acute stroke

DETAILED DESCRIPTION:
The study will include a Screening/Baseline Period, a Treatment Period, and a Post-treatment Follow-up Period. During the Screening Period, subjects will be selected for the study on the basis of inclusion and exclusion criteria (see below). A screening computed tomography scan to exclude brain bleeding will be performed. The patient's informed consent will be obtained. The patient will be randomly allocated to DP-b99 or placebo. Immediately after this randomization and baseline assessments (lab tests and ECG), subjects will be given a 2-hour intra-venous infusion of DP-b99 or placebo. Additional 3 such infusions will then be given daily to a total of 4 consecutive treatment days, which make up the "Treatment Period". Throughout the 4-day Treatment Period the treatment's safety and the National Institutes of Health Stroke Scale (NIHSS) score will be evaluated daily. (The NIHSS assesses certain abilities of the patient, e.g. strength, speech, vision and coordination). If their condition requires, patients may have to stay in hospital more than these 4 days, regardless of their participation in the study.Subjects will be further assessed for NIHSS score changes and safety (lab tests and ECG) during the Post-treatment Follow-up Period, with data collected 30 and 90 days after the stroke. Other outcome scales (Barthel Index and Modified Rankin Scale) will be also used in the Day 30 and Day 90 visits

ELIGIBILITY:
Patients that may enter the study:

* Patients with ischemic stroke, (that is, stroke that results from a blockage of blood flow to part of the brain), which is accompanied by language dysfunction (e.g. inability to understand speech), visual field defect or inattention to one side of the body or the space around the patient.
* Patients in whom the study treatment can start no less than 1 and not more than 9 hours after the stroke's onset
* Patients with moderate-severe degree of neurological deficit in the 9 hours after stroke onset (defined as NIHSS score of 7 to 20
* Patients that can understand the requirements of the study and are willing to provide written informed consent (If the subject is incapacitated, informed consent will be sought from a legally acceptable representative.)

Patients that cannot participate:

* Patients with a brain (intracerebral or subarachnoid) hemorrhage per screening computed tomography scan candidates for thrombolytic therapy for the current stroke patients having a mental impairment that renders them incapable to understand the study's requirements patients with other diseases that in the investigator's opinion may lead, independently of the current stroke, to further deterioration in the subject's neurological status during the trial period, or may confuse the evaluation of the present stroke
* Patients likely to undergo a procedure involving cardiopulmonary bypass during the study period
* Patients with medical conditions that may not enable them to complete the study (e.g life-threatening diseases,)
* Patients whose condition improves already during the screening period
* Patients who already have functional limitations before the present study (retrospective Modified Rankin Scale score of >3)
* Patients who suffered a stroke within the past 90 days that seems to have been in the same brain region as the current acute stroke
* Patients with severe hypertension (systolic BP >210 mm Hg or diastolic BP >120 mm Hg) or hypotension (systolic BP <90 mm Hg), Patients with significant history of renal or liver disease(s) (serum creatinine of > 2.0 mg/dL; alanine aminotransferase, aspartate aminotransferase, or gamma-glutamyl transferase values of > threefold the upper normal limit)
* Patients with a platelet count of <100,000/mm3
* Female patients of childbearing potential who are not using adequate and effective birth control measures or who are pregnant or lactating (the screening evaluation of female subjects of childbearing potential will include a serum pregnancy test.)
* Patients who are users of addictive agents, or alcoholics
* Patients who have received an investigational drug within the 90 days before the present stroke or such that are past recipients of DP-b99

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-02; Study Completion 2006-10

PRIMARY OUTCOMES:
Change in the National Institutes of Health Stroke Scale (NIHSS) score from baseline to Day 90

SECONDARY OUTCOMES:
Safety and tolerability Neurological recovery and function

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Rosenberg, M.D., Study Director — D-Pharm Ltd.
Locations (22):
- Germany (17):
  - Neurologische Klink GmbH der Rhoen-Klinikum AG, Bad Neustadt / Saale
  - Charité - Universitätsmedizin Berlin / Campus Charité Mitte, Klinik und Poliklinik für Neurologie, Berlin
  - Klinik und Poliklinik für Neurologie Klinikum der Universität zu Köln, Cologne
  - Universitätsklinik Essen Klinik und Poliklinik für Neurologie, Essen
  - Neurologische Universitätsklinik Abteilung für Neurologie, Freiburg im Breisgau
  - Universitätsklinikum Leipzig Klinik und Poliklinik für Neurologie, Leipzig
  - Otto-von-Guericke-Universität Magdeburg Medizinische Fakultät, Klinik für Neurologie, Magdeburg
  - Johannes Gutenberg-Universität Mainz Neurologische Klinik, Mainz
  - Klinikum 1 Minden Neurologische Klinik, Minden
  - Neurologische Klinik und Poliklinik Technische Universität München Klinikum rechts der Isar, München
  - Städtisches Krankenhaus München-Bogenhausen Abteilung für Neurologie und Klinische, München
  - Städtisches Krankenhaus München-Harlaching Abteilung für Neurologie, München-Harlaching
  - Universitätsklinikum Münster Klinik und Poliklinik für Neurologie, Münster
  - Klinikum Osnabrück Abteilung Neurologie, Osnabrück
  - Knappschaftskrankenhaus Recklinghausen Klinik für Neurologie und Klinische Neurophysiologie, Recklinghausen
  - Universitätsklinikum Ulm Abteilung für Neurologie im RKU, Ulm
  - Medizinisches Zentrum Kreis Aachen gGmbH Klinik für Neurologie, Würselen-Bardenberg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Result] Oral Session on Acute stroke: treatment concepts, presented on Thursday, 31 May 2007 at the XVI. European Stroke Conference, Glasgow, United Kingdom, 29 May - 1 June 2007. The abstract can be found at: http://www.esc-archive.eu/glasgow07/gla_so10_1.asp
- See also: Click here for more information on the sponsor — http://www.dpharm.com